CLINICAL TRIAL: NCT05115708
Title: Kahook Dual Blade Ab-interno Trabeculotomy Versus ab Externo Viscotrabeculotomy in Primary Congenital Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Mohammed Elsayed Abdelkader, Assisstant professor of ophthalmology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R.21.10.1477
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Glaucoma; Congenital Glaucoma
MeSH Terms: conditions — Glaucoma; Hydrophthalmos

STUDY DESIGN:
Intervention Model Description: Kahook dual blade ab-interno Trabeculotomy versus ab externo viscotrabeculotomy in treatment of primary congenital glaucoma.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kahook dual blade ab-interno Trabeculotomy (Active Comparator): The Kahook dual blade® (KDB) assisted ab-interno trabeculotomy
  Interventions: Procedure: The Kahook dual blade® (KDB) assisted ab-interno trabeculotomy
- ab externo viscotrabeculotomy (Active Comparator): In brief, a fornix-based conjunctival incision is followed by fashioning and dissection of a triangular scleral flap. Radial incisions at the limbus followed to identify Schlemm's canal. viscotrabeculotomy, is performed by injection of high-viscosity sodium hyaluronate (Healon GV, Pfizer, NY) into Schlemm's canal prior to completion of the procedure with the metal trabeculotome. while a Nylon 10/0 suture in inserted into schlemm's canal in visco-circumferential-suture trabeculotomy group.
  Interventions: Procedure: ab externo viscotrabeculotomy

INTERVENTIONS:
Procedure: ab externo viscotrabeculotomy — In brief, a fornix-based conjunctival incision is followed by fashioning and dissection of a triangular scleral flap. Radial incisions at the limbus followed to identify Schlemm's canal. viscotrabeculotomy, is performed by injection of high-viscosity sodium hyaluronate (Healon GV, Pfizer, NY) into Schlemm's canal prior to completion of the procedure with the metal trabeculotome. while a Nylon 10/0 suture in inserted into schlemm's canal in visco-circumferential-suture trabeculotomy group
  Arms: ab externo viscotrabeculotomy
Procedure: The Kahook dual blade® (KDB) assisted ab-interno trabeculotomy — The Kahook dual blade® (KDB) assisted ab-interno trabeculotomy
  Arms: Kahook dual blade ab-interno Trabeculotomy

SUMMARY:
This prospective study aims to compare KDB ab-interno trabeculotomy to ab externo rigid probe viscotrabeculotomy in patients with PCG.

DETAILED DESCRIPTION:
Introduction:

Ab externo viscotrabeculotomy is known as an effective surgical procedure used for managing primary congenital glaucoma (PCG) in which the Schlemm's canal (SC) is identified and a metal probe is inserted into the canal and rotated into the anterior chamber (AC) to perforate the SC inner wall.

Recently, Kahook dual blade (KDB) have been developed as one of the micro-invasive glaucoma surgical tools which removes a strip of the trabecular meshwork(TM) at the angle with superiority to simple goniotomy in treating the angle pathology in PCG.

The Kahook dual blade® (KDB) assisted ab-interno trabeculotomy is a simple procedure usually performed at the time of cataract surgery. It doesn't require sutures, and it carries no risk of bleb leaks or infections. It has a a quicker postoperative visual recovery than most other glaucoma treatments. The KDB device is specifically designed to produce targeted and fine tuned parallel incisions in the trabecular meshwork tissue for a quick and effective glaucoma treatment. The KDB's unique design enables precise excision of diseased trabecular meshwork (TM) to access multiple collector channels.

The KDB's unique design enables the operator to perform excisional goniotomy both during cataract surgery and as a stand alone procedure. The Kahook Dual Blade is a precise, intuitive surgical instrument utilized to perform excisional goniotomy.

Purpose:

This prospective study aims to compare KDB ab-interno trabeculotomy to ab externo rigid probe viscotrabeculotomy in patients with PCG.

Methods:

Sixty eyes of with PCG underwent ab-interno trabeculotomy using a KDB or ab externo viscotrabeculotomy. The study will be conducted at Mansoura university ophthalmic Center. Follow-up visits were scheduled at these post-operative dates: first day, first week, first month, 3rd month and then every 3 months for 2 years. Complete success was defined as an IOP from 6 to 17 mmHg at the 2-year follow-up visit, without AGM or further surgical interventions, without any sign of glaucoma progression (increasing corneal diameter, axial length or cup/disc ratio) and without visual devastating complications. Qualified success was defined as fulfilling the same criteria but with the use of AGM.

Preoperative data including age, sex, laterality, type of glaucoma, ocular history, number of glaucoma medications, IOP, cup to disc ratio, and central corneal thickness (CCT) were record. Postoperative data included follow-up durations.

Statistical analysis:

All statistical analysis will be accomplished using IBM SPSS version 20. Assessment of the data normality will be done using both Histogram plot and Shapiro-Wilk's test. Wilcoxon test was used to compare the preoperative and postoperative variables in each group. The comparison between the two groups will be done using Mann-Whitney test for numerical variables and Chi-square test for categorical variables. Kaplan-Meier survival curve will be plotted to estimate the mean survival time and probabilities of failure at different follow-up stages in the both groups. For all tests, P value of less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

primary congenital glaucoma

Exclusion Criteria:

secondary congenital glaucoma

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
IOP | 2 years
  Complete success was defined as an IOP from 6 to 17 mmHg at the 2-year follow-up visit, without AGM or further surgical interventions, without any sign of glaucoma progression (increasing corneal diameter, axial length or cup/disc ratio) and without visual devastating complications. Qualified success was defined as fulfilling the same criteria but with the use of AGM.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Elwehidy, DM, Study Chair — Mansoura faculty of medicine
Locations (1):
- Mansoura university ophthalmic center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
share primitive data as supplementary digital content
Supporting Information: Study Protocol, SAP, ICF